# The Cleveland Clinic Consent to Participate in a Research Study

# **ANCILLARY EFFECTS OF ORAL NALOXEGOL (MOVANTIK)**

Principal Investigator:Dr. Alparslan Turan, MD(216) 445-9857Study Coordinator:Steve Leung, MD(216)-636-5493After hours phone contact #:CCF Page Operator(216) 444-2200

You are being invited to participate in a research study. A research study is designed to answer specific questions about new ways to prevent, detect, and treat disease. Being in a research study is different from being a patient. The purpose of this document is to provide a written summary of the discussion and exchange of research information you had with the research team. It is also for use as a reference during the study.

#### Please note:

- You are being asked to participate in a research study.
- Ask as many questions as needed so you can make an informed decision.
- Carefully consider the risks, benefits, and alternatives of the research.
- Your decision to participate is completely voluntary and will have no effect on the quality of your medical care if you choose not to participate. You can also withdraw from the study at anytime.

This research study has been approved by the Institutional Review Board (IRB). The IRB is a committee that reviews human research studies to ensure that the safety and welfare of research volunteers are protected in accordance with federal human subject regulations and ethical principles.

#### 1. INFORMATION ON THE RESEARCH

### Why is the research study being done?

The purpose of this study is to find out whether oral Naloxegol can reduce the side effects of opioid painkillers following surgery. Opioids are the gold standard for postoperative pain management, but they have been shown to produce uncomfortable side effects such as urinary retention (an inability to completely empty the bladder), constipation and nausea/vomiting. Clinical evidence demonstrates that Naloxegol can safely and effectively block these undesirable side effects while maintaining the painkilling effects of opioids in outpatients suffering from opioid-induced constipation. This study aims to explore whether Naloxegol can similarly reduce opioid-induced side effects in post-surgical patients. About 130 surgery patients will participate in this study which is being conducted at Cleveland Clinic Main Campus. As a patient who is undergoing elective surgery at Cleveland Clinic, you are being invited to participate in this research study.

### What is involved if you decide to take part in this research study?

If you agree to participate in this study, you will be randomly placed into one of two treatment groups: Naloxegol or placebo. Neither the study team nor you as the study participant can choose which group you are in. Your group assignment is chosen by chance – like the flip of a coin. You have an equal chance of being assigned to either treatment group.

Participants in the Naloxegol group will be given the investigational drug, an oral tablet, on the morning of surgery as well as on post-operative days 1, 2 and 3. Participants in the placebo group will receive an oral tablet that is equal in size, shape and color to the investigational drug according to the same time schedule. Only the Pharmacy team will have access to which participants are in which group in the event of a safety or emergency situation.

For both treatment groups, all intraoperative and postoperative pain medications will be left to the discretion of the staff anesthesiologist.

You will also be asked to participate in the following study procedures:

#### Bladder Scans

Opioid-induced urine retention is a common side effect for patients, and it is our primary outcome measure in this study. Therefore we will use a portable Bladder Scan<sup>TM</sup> BVI 3000<sup>®</sup> to measure the volume of urine that remains in the bladder following urination. The scanner will be placed above the pubic area and held stationary during measurement of bladder diameter as well as residual urine volume. Bladder scans take approximately 5 minutes and will be performed by trained MD research fellows twice per day on postoperative days 1, 2 and 3.

## Surveys/Questionnaires

You will be asked to provide information about your social and medical history including but not limited to tobacco use, kidney disease, diabetes mellitus, chronic pain conditions, etc. You will also be asked to complete the following questionnaires:

<u>Opioid-Related Symptom Distress Scale</u> – you will be asked about frequency, severity and discomfort for 12 opioid-related side effects

<u>Opioid Complications Survey</u> – you will be asked about complications such as nausea, vomiting, itching, etc.

<u>Myles Quality of Recovery Scale</u> – you will be asked about your early postoperative health status.

<u>Patient Satisfaction Survey</u> – you will be asked at discharge about your satisfaction with your recovery.

Lastly, you will be asked to let the study team collect demographic and clinical information from your electronic medical record throughout your enrollment in the study including but not limited to:

- Height, weight, age, ethnicity, etc.
- Preoperative laboratory results and medications
- Intraoperative opioid consumption, operation time and surgery type
- Postoperative opioid consumption, side effects and laboratory data
- Functionality such as bathing, toileting, walking and moving

Participation in this study will end on post-operative day 3 or the day you are discharged from the hospital, whichever comes first.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U. S. law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search the Website at any time.

#### 2. ALTERNATIVES

### What are the alternatives to participation in the research study?

Agreeing to participate in this research will not change the normal medical care which you are receiving. Your alternatives are to participate in this research or not to participate in this research, but this will change nothing about your medical care.

#### 3. RISKS

### What are the risks of participating in the research study?

More Common: >10%

• Abdominal pain

Common: 1% to 10%

- Nausea
- Diarrhea
- Headache
- Vomiting
- Flatulence
- Hyperhidrosis
- Nasopharyngitis (Respiratory)

There may be unforeseen risks to an unborn child associated with taking Naloxegol. Therefore, if you are capable of giving birth to or fathering a child, you and your sexual partner should use adequate birth control measures while you are in the study. These measures may include abstinence, oral contraceptives (birth control pills), IUD, diaphragm, approved hormone injections, condoms, or documentation of medical sterilization. If you are unwilling to do this, we ask that you do not participate in this study.

Pregnancy tests will be performed on all women of child-bearing potential before beginning the study. If you or your spouse becomes pregnant while taking part in this study, you must notify the study doctor immediately.

#### 4. BENEFITS

## What are possible benefits of participating in the research?

Participation in this research study may or may not reduce the unpleasant side effects of opioid use; however the knowledge to be gained may benefit surgical patients in the future.

#### 5. COSTS

### Are there any costs to you if you participate in this study?

Some of the services you will receive during this research study are considered to be conventional routine clinical services that you would have received even if you were not participating in the research study and will be billed to you or your health insurance plan. Examples of these routine services include your surgical procedure and all related tests, labs and images. You are responsible for paying any deductibles, co-payments or co-insurance that are a normal part of your health insurance plan.

The following research study services are being done only because you are participating in this research study and **will be paid for by the study sponsor** and will not be billed to you or your health insurance plan. These "research only" services include: study drug or placebo and all bladder scans.

#### 6. COMPENSATION

### Are there any payments to you if you participate in this study?

There is no financial compensation for participating in this study.

### What happens if I am injured as a result of participation in this research?

In the event you are injured as a result of participation in this research, medical care is available to you. The costs of such medical care will be billed to you or your insurance company. There are no plans to provide compensation for lost wages, direct or indirect losses. The Cleveland Clinic will not voluntarily provide compensation for research related injury. You are not waiving any legal rights by signing this form. Further information about research related injury is available by contacting the Institutional Review Board at (216) 444-2924.

### 7. PRIVACY AND CONFIDENTIALITY

# What will happen to your information that is collected for this research?

Cleveland Clinic has rules and procedures to protect information about you. Federal and State laws also protect your privacy.

The research team working on the study will collect information about you. This includes your health information, data collected for this research study, and personal identifying information including your name, address, date of birth and other identifying information.

Generally, only people on the research team will know your identity and that you are in the research study. However, sometimes other people at Cleveland Clinic may see or give out your information. These include people who review research studies including the Institutional Review Board and Research Compliance, their staff, lawyers, or other Cleveland Clinic staff.

People outside Cleveland Clinic may need to see your information for this study. Examples include government groups (such as the Food and Drug Administration), safety monitors, other hospitals in the study, and the sponsor of the research and their agents. As Cleveland Clinic we will do our best to ensure your information is kept confidential and that only

the health information which is minimally required to conduct the study is used or disclosed to people outside Cleveland Clinic; however, people outside Cleveland Clinic who receive your information may not be covered by this promise.

You do not have to give this permission to use and give out your information; however you will not be able to participate in this research study without providing this permission by signing this consent form. The use and disclosure of your information has no expiration date.

You may cancel your permission to use and disclose your information at any time by notifying the Principal Investigator in writing: Dr. Alparslan Turan, at the Cleveland Clinic, 9500 Euclid Avenue/P77, Cleveland, Ohio 44195. If you do cancel your permission to use and disclose your information, your participation in this study will end, and no further information about you will be collected. However, your cancellation would not affect information already collected in the study.

The results of this study will not be directly shared with participants, however any research that is published as a result of our findings will preserve the confidentiality of all participants and is accessible to the general public.

#### 8. CONFLICT OF INTEREST

### Do the researchers or institution have any conflicts of interest relating to this study?

One or more of the Investigators conducting this study may serve as paid speakers, consultants to advisory committee members for the company that is paying for this research or a company that makes products used in this study. These financial interests are within permissible limits established by the Cleveland Clinic Conflict of Interest Policy. If you have any questions, please ask your study doctor or call the Institutional Review Board at (216) 444-2924.

### 9. QUESTIONS

### Who do you call if you have any questions or problems?

If you have any questions or concerns about the research or develop a research-related problem, you should contact Dr. Alparslan Turan at 216-445-9857 or Steve Leung at 216-636-5493 during business hours or via the CCF operator (216) 444-2200 after business hours. If you have any questions about your rights as a research subject, you should contact the Institutional Review Board at (216) 444-2924.

#### 10. VOLUNTARY PARTICIPATION

#### What are your rights as a research participant?

Taking part in this study is voluntary. You will be told of any new, relevant information from the research that may affect your health, welfare, or willingness to continue in this study. You may choose not to take part or may leave the study at any time. Withdrawing from the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to

withdraw from the study you should discuss with your study doctor your decision to ensure a safe withdrawal.

#### 11. SIGNATURES

### **Statement of Participant**

I have read and have had verbally explained to me the above information and have had all my questions answered to my satisfaction. I understand that my participation is voluntary and that I may stop my participation in the study at any time. Signing this form does not waive any of my legal rights. I understand that a copy of this consent will be provided to me. By signing below, I agree to take part in this research study.

Printed name of participant

Participant Signature

Date

Statement of Person Conducting Informed Consent Discussion

I have discussed the information contained in this document with the participant and it is my opinion that the participant understands the risks, benefits, alternatives and procedures involved with this research study.

Printed name of person obtaining consent

Date

Signature of person obtaining consent